CLINICAL TRIAL: NCT06166407
Title: The Breisgau Pheno Heart Study
Brief Title: Breisgau Pheno Heart Study
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Patrick Siegel, MD, University Hospital Freiburg
Other Study IDs: BPHS
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Myocardial Infarction; STEMI; NSTEMI
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Coronary heart disease and its acute complication, myocardial infarction (MI), represent the leading causes of death in Europe and the United States. Although novel treatment strategies have helped to improve survival in patients with MI, a large proportion of patients develops heart failure and is at risk of life-threatening arrhythmias. Complications arising after MI constitute a severe burden not only for the patients themselves, but also for health care systems worldwide.

The likelihood of these complications depends on the area of myocardial tissue lost and the process of myocardial repair and scar tissue formation after MI ('remodeling') which are modified by the local and systemic immune response after MI. The immune response is critical after myocardial infarction. In particular, sustained overactive and prolonged inflammatory reactions lead to accentuated myocardial damage and dysfunction. Important mediators of the inflammatory reaction after MI are monocytes, T-cells, B-cells and hematopoietic stem and progenitor cells. Following MI, myeloid cells derived from the hematopoietic system drive a sharp increase in systemic leukocyte levels that correlates closely with mortality. T- and B-cells in particular act in response to specific antigens. Most of the data regarding the inflammatory response after MI, however, are derived from animal models. The immunological phenotypes after MI and their association with clinical outcome in humans are insufficiently characterized.

Aims: The aim of this project is to provide establish clinically and immunologically well-characterized cohort of patients after MI This will aid in identifying novel prognostic cellular and humoral biomarkers that may be used to identify patients at a high inflammatory and immune risk and to guide clinical management. Furthermore, these mediators, in the future, may be targeted by novel antigen-specific immunomodulatory approaches.

Patients with myocardial infarction (STEMI and NSTEMI) will be recruited after PCI within 24h and receive a structured follow-up. Clinical read-outs include a detailed and standardized patient history, clinical examination, standard blood work, coronary angiography, ECG, echocardiography and for subgroups, MRI. Patients will present for study visits at 6 weeks, 3 months and 12 months after the initial event. Blood will be sampled at the inclusion and during follow-up visits. Peripheral blood mononuclear cells and plasma will be stored at the Cardiovascular BioBank (CVBB) and FREEZE, both institutions at the University Hospital in Freiburg. Major adverse cardiac events (myocardial infarction, stroke, hospitalization for heart failure, cardiovascular death) will be recorded using telephone interviews and standardized queries to the local authorities. Several laboratory read-outs are planned including flow cytometry, mass cytometry, single cell RNA sequencing, T cell and B cell receptor sequencing and bulk-RNA-sequencing. In an initial approach we aim to recruit 400 patients with MI, of which we expect ≈40 to develop ischemic cardiomyopathy. Differences in immunological profiles between patients that develop MI and a propensity-matched control group will then be analyzed and correlated with clinical outcome data.

ELIGIBILITY:
Inclusion Criteria:

* Emergency coronary angiography and age>18 years and STEMI or NSTEMI or "none of these diseases"

Exclusion Criteria:

* Hemoglobin<7,0 g/dl
* Platelets <50.000/µl
* Unable to provide written informed consent
* Age > 80 years
* hematological neoplasia
* metastasized cancers
* acute infection (z.B. Sepsis)
* Chronic Inflammatory conditions (z.B. inflammatory bowel disease, Rheumatoid arthritis, chronisch hepatitis)
* Pregnancy
* Immunosuppression
* Resuscitation >5 min oder mehr als 1x Defibrillation vor Koronarangiographie
* Cardiogenic shock
* Mechanical circulatory support
* Cardiomyopathy with an left ventricular ejection fraction F <40% before the event
* Dialysis
* Cirrhosis > CHILD-A
* Not living in the county of Breisgau-Hochschwarzwald or Emmendingen oder planned relocation
* Alcohol and drug abuse
* Non-compliance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with STEMI and NSTEMI
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | years
  composite endpoint of Stroke, MI, hospitalization for heart failure, cardiovascular death, revascularization

SECONDARY OUTCOMES:
Diagnosis of atrial fibrillation | years
  Atrial fibrillation diagnosis by 12-lead ECG

IPD SHARING:
Plan to Share IPD: No